CLINICAL TRIAL: NCT04258657
Title: Neoadjuvant Chomotherapy With Paclitaxel-albumin and S-1 for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-GCCT
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel-albumin and S-1 (Experimental)
  Interventions: Drug: paclitaxel-albumin and S-1

INTERVENTIONS:
Drug: paclitaxel-albumin and S-1 — neoadjuvant chomotherapy with paclitaxel-albumin and S-1 for advanced gastric cancer

SUMMARY:
This is a interventional clinical trial to assess the efficacy and safety of combinational therapy of paclitaxel-albumin and S-1 for the neoadjuvant chemotherapy of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed gastric adenocarcinoma
2. Type II and III esophageal-gastric-junction malignancy
3. AJCC stage II-III
4. No contraindications for surgery, radical resection can be expected
5. KPS>60; ECOG score:0-2
6. Expactant survival period>6 months
7. Age 20~75
8. No other major health issues
9. Lab results within 7 days before inclusion must satisfy:

   1. neutrophil≥1.5×109/L
   2. PLT≥100×109/L
   3. hemogloblin≥90g/L
   4. ALT,AST<1.5 upper limit
   5. Tbil≤1.0×UNL
   6. serum creatinine<1.5×UNL
   7. PT-INR/PTT<1.7 upper limit
10. with measurable lesion according to RECIST1.1 criteria
11. with consent
12. co-operative

Exclusion Criteria:

1. with other major health issue
2. allergic to relevant drugs
3. experienced any other drug therapy with 4 weeks before inclusion
4. experienced any drug therapy for gastric cancer at anytime
5. diagnosed with any other malignancy within the past 5 years
6. women at child-bearing age; pregnant or breast-feeding women
7. with severe heart disease
8. with upper GI digestion or disrupted absorption
9. with peripheral neural disease
10. with transplated organs or organs having been resected for transplantation
11. known DPD deficiency
12. with uncontrolled infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 3-year
  disease free survival

SECONDARY OUTCOMES:
ORR | 3-year
  objective response rate
OS | 3-year
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, Study Director — Beijing Friendship Hospital
Locations (1):
- Zhongtao Zhang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided